CLINICAL TRIAL: NCT07249567
Title: Comparison of Respiratory and Peripheral Muscle Strength, Exercise Capacity, and Muscle Oxygenation in Individuals With COPD and PRISM
Brief Title: Comparison of Patients With COPD and PRISM
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-2383
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with COPD: Patients with chronic obstructive pulmonary disease will be included.
- Patients with PRISm: Patients with preserved ratio impaired spirometry will be included.
- Control: Healthy controls will be included.

SUMMARY:
COPD is a preventable and treatable lung disease characterized by persistent and progressive airflow limitation. PRISm, on the other hand, is a spirometry pattern that does not meet COPD diagnostic criteria despite symptoms and functional impairments, but requires maintenance. PRISm can predispose to the development of COPD and exacerbations, and can reduce exercise capacity by reducing respiratory function and oxygen consumption. There are no studies in the literature comparing respiratory muscle strength, peripheral muscle strength, and oxygenation in PRISm, COPD, and healthy individuals. Therefore, this study aimed to evaluate these parameters and compare them with healthy individuals.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common, preventable, and treatable multisystem lung disease characterized by chronic respiratory symptoms (dyspnea, cough, sputum production, and/or exacerbations) due to airway abnormalities, causing persistent and often progressive airflow limitation. PRISm is defined as a spirometry pattern that is not always a stable phenotype but should be considered "sick" because symptoms and/or functional and/or structural abnormalities are present and therefore require care and treatment. Recently, PRISm has been identified as a subtype more prone to developing COPD or experiencing acute exacerbations. In addition to affecting the respiratory muscles, PRISm's effects on respiratory function lead to decreased body oxygen consumption and increased dyspnea. PRISm can also lead to decreased exercise capacity due to the respiratory problems and dyspnea it causes. Although there are not enough studies in the literature investigating exercise capacity and lung functions on behalf of PRISm, no previous study comparing respiratory muscle strength, peripheral muscle strength and oxygenation in PRISm, COPD and healthy individuals has been found.

ELIGIBILITY:
Inclusion Criteria:

For the COPD group:

* Being >40 years old,
* Being diagnosed with COPD,
* Being clinically stable,
* Volunteering to participate in the study.

For the PRISm group:

* Being >40 years old,
* Being diagnosed with PRISm,
* Volunteering to participate in the study.

For the healthy control group:

* Being >40 years old,
* Volunteering to participate in the study.

Exclusion Criteria:

For the COPD group:

* Having severe orthopedic, neurological, or cardiac diseases,
* Being in a COPD exacerbation,
* Having a comorbid lung disease,
* Being on clinically unstable medication,
* Voluntarily not participating in the study.

For the PRISm group:

* Being diagnosed with COPD,
* Having severe orthopedic, neurological, or cardiac diseases,
* Having a comorbid lung disease,
* Voluntarily not participating in the study.

For the healthy control group:

* Having a known chronic disease,
* Voluntarily not participating in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD and PRSIm will be included and compared with healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | Baseline
  Upper extremity exercise capacity will be evaluated with the six-minute pegboard and ring test (6-PBRT).
Lower extremity exercise capacity | Baseline
  Lower extremity exercise capacity will be evaluated with six- minute walking test.
Peripheral muscle strength | Baseline
  Peripheral muscle strength will be evaluated with a dynamometer.
Muscle oxygenation | Baseline
  Muscle oxygenation assessment will be performed using the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA).
Respiratory Muscle Strength | Baseline
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be evaluated.
Respiratory Muscle Endurance | Baseline
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load.
Dyspnea | Baseline
  Dyspnea is assessed with the modified Medical Research Council (mMRC) dyspnea scale. As the score increases, shortness of breath increases.
Clinical symptoms | Baseline
  The COPD Assessment Test will be evaluated. This scale scored on a 0-5 point scale to assess symptoms associated with COPD. As the score increases, the symptom increases.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity (FVC) | Baseline
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced vital capacity (FVC) will be measured.
Pulmonary function (Forced expiratory volume in the first second (FEV1) | Baseline
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (FEV1 / FVC) | Baseline
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. FEV1 / FVC will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Baseline
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Pulmonary function (Peak flow rate (PEF)) | Baseline
  Pulmonary function will be evaluated using the spirometry, according to American Thoracic Society and European Respiratory Society criteria. Peak flow rate (PEF) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Güneş, PhD, Principal Investigator — Karabuk University; Rabia Hande Avcı, MD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No